CLINICAL TRIAL: NCT06887556
Title: Mpox Comprehensive Assessment for Responsive Immunisation in Emergency Outbreaks
Acronym: MPOX CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Rwanda Biomedical Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Mpox CARE
Record Dates: First submitted 2025-02-18; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-11

CONDITIONS: Mpox
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): All participants will receive the same interventions.
  Interventions: Diagnostic Test: ELISA; Diagnostic Test: Lateral flow assay

INTERVENTIONS:
Diagnostic Test: ELISA — Mpox-specific antibody ELISA
Diagnostic Test: Lateral flow assay — Dried blood spot lateral flow assay for Mpox antibody

SUMMARY:
The MPXV CARE study principally aims to use clinical and epidemiology data to target specific individuals willing and able to provide appropriate and proportionate biological samples to develop novel immune diagnostics that support models of disease burden and future vaccine utilisation.

DETAILED DESCRIPTION:
Cases of Mpox in Central and East Africa have been climbing since December 2022 when Democratic Republic of Congo (DRC) declared a national outbreak of the disease. There are two strains of circulating virus, clade Ia (previously known as clade I) in northwestern DRC primarily affecting children, and a new strain clade Ib in northeastern DRC which has since spread to bordering countries. The clade Ib strain, sub-lineage A was first identified in South Kivu. This strain has been found to have a APOBEC3-type mutations allowing increased circulation between humans. This novel clade is mainly characterized by the gene insertions and deletions including the deletion on C3L gene that effect the CDC recommended Clade I-specific real-time PCR detection. The WHO Director General declared the outbreak a public health emergency on 14th August 202433 as a result of escalating case numbers of both clade I strains. As of 28July 2024, this year there have been a total of 14,250 cases in 10 African countries, with a case fatality of 3.2%. This is likely to be an underestimate given the limited testing and healthcare capacity in some of the regions affected. The clade 1b Mpox outbreak is an urgent public health emergency in need of scientific countermeasures to control the spread of disease and protect African communities.

The primary clinical aim of this study to develop novel immune diagnostics to estimate Mpox's sero-prevalence and determine exposure to Mpox virus and/or previous vaccination as a tool for vaccine prioritization among at risk populations.

Participants will be recruited from the following groups:

* Group 1 (suspected exposure cohort): asymptomatic volunteers at risk of Mpox including:

  * Those who live within or adjacent to, or spend prolonged amounts of time in an epidemiologically identified region of Mpox transmission
  * Close contacts of those with microbiologically confirmed Mpox
* Group 2 (post-exposure/vaccinated cohort):

  * asymptomatic volunteers who have had clinically or microbiologically confirmed Mpox infection within the last one-month (group 2a) or more than one-month ago (group 2b)
  * Those who have received a smallpox/MVA vaccine within the last one-month (group 2c) or more than one-month ago (group 2d)
* Group 3 (control cohort): asymptomatic volunteers with no known exposure to Mpox

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females aged between ages 5-80 years, who are able and willing to provide informed consent and will comply with the study requirements.
* Group 1 (suspected exposure cohort) only

  * Live within or adjacent to an epidemiologically identified region of Mpox transmission
  * Close contacts of those with microbiologically confirmed Mpox
* Group 2 (post-exposure/vaccinated cohort) only

  * Previous clinically or microbiologically confirmed Mpox or confirmed previous vaccination with a smallpox/MVA vaccine
  * Fully recovered from Mpox infection
* Group 3 (control cohort) only:

  * Asymptomatic with no known exposure to Mpox

Exclusion Criteria:

* Unwilling or unable to provide informed consent to take part
* Unwilling or unable to comply with study procedures
* History of any suspected or confirmed disorder of the immune system that, in the opinion of the investigators, might impair the results of the study
* Have a bleeding disorder deemed significant by a member of the study team
* Pregnant or breast-feeding females
* Group 1 (suspected exposure cohort) only

  * Known history of Mpox infection
  * Current symptoms consistent with Mpox
  * Known exposure to Mpox in the last month
* Group 2 (post-exposure/vaccinated cohort) only

  * Participants with any ongoing symptoms of Mpox, indicating incomplete recovery.
* Group 3 (control cohort only)

  * Symptoms of Mpox
  * Known exposure to Mpox in the last month

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Detection of anti-Mpox specific IgG antibody by ELISA | Day 1
  Number of patients in whom anti-Mpox specific IgG antibody is detected
The clinical diagnostic performance of the RDT for Mpox exposure confirmation | Day 1
  A blood sample will be tested on the lateral flow device which will give a positive/negative result for the presence of antibody. This will be compared to the gold standard testing modality of ELISA. The MPox POC LFT performance versus ELISA will be characterised by test sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and likelihood ratios.

SECONDARY OUTCOMES:
Perspectives of healthcare workers and the public on studies in response to outbreaks | Day 1
  Qualitative analysis of output from focus group discussion regarding taking part in this trial
Perspectives of healthcare workers and the public on the development of novel immune diagnostic tools | Day 1
  Qualitative analysis of focus groups with the healthcare workers and the public who have taken part in the study around this topic.
Perspectives of healthcare workers and the public on the vaccine cold-chain readiness to support public health measures | Day 1
  Qualitative analysis of focus groups with the healthcare workers and the public who have taken part in the study around this topic.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Green, Principal Investigator — University of Birmingham
Locations (1):
- Rwanda Biomedical Center, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are not openly available to protect the confidentiality of study participants. Fully anonymised data are, however, available from the authors upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting immediately after article publication and the data will be made accessible for up to 5 years. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a methodologically sound research proposal. Data must be required to achieve the aims in the approved proposal. Data requests should be directed to c.a.green.2@bham.ac.uk.